CLINICAL TRIAL: NCT05915598
Title: Investigating the Effects of Right/Left Discrimination Training on Pain Perception and Functional Disability in Fibromyalgia Patients: A Randomized Controlled Trial
Brief Title: Right/Left Discrimination Training on Fibromyalgia Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/0059000012
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Right/left discrimination training: The training program will consist of tasks such as identifying the laterality of images (e.g., hands, feet, faces) and sounds (e.g., spatially localized sounds). The tasks will be designed with increasing levels of difficulty to challenge participants and promote skill development.
  Training schedule: Participants will be instructed to engage in the right/left discrimination training for 20 minutes per day, 5 days per week, over a six-week period. They will be encouraged to complete the training sessions at consistent times to support habit formation.
  Monitoring and feedback: The research team will remotely monitor participants' progress and provide personalized feedback on a weekly basis. This will include reviewing performance metrics within the app, discussing any challenges or barriers to adherence, and offering guidance to support continued engagement in the training program.
  Interventions: Other: Right/left discrimination training
- Control group (Active Comparator): Usual care: Participants will continue their usual care management for fibromyalgia, including any prescribed medications and physician consultations. No specific right/left discrimination training will be provided to the control group.
  Interventions: Other: usual care

INTERVENTIONS:
Other: Right/left discrimination training — Participants will use recognize app by Neuro-orthopedic institute (NOI) for daily right/left discrimination training.
  The training will include visual and auditory stimuli, with tasks such as identifying the laterality of images and sounds.
  Participants will engage in training for 20 minutes per day, 5 days per week, over a six-week period.
  Weekly monitoring and feedback will be provided by the research team
  Arms: Intervention group
Other: usual care — Usual care: Participants will continue their usual care management for fibromyalgia, including any prescribed medications and physician consultations. No specific right/left discrimination training will be provided to the control group.
  Follow-up assessments: Participants in the control group will undergo the same follow-up assessments as the intervention group to evaluate changes in pain perception, functional disability, and cognitive function.
  Arms: Control group

SUMMARY:
To determine whether a targeted right/left discrimination training program can improve pain perception and functional disability in fibromyalgia patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia according to the 2016 American College of Rheumatology criteria
* Adults between 35 - 55 years old
* Both sexes
* Stable medication use for at least one month prior to enrollment

Exclusion Criteria:

* History of other musculoskeletal or neurological disorders
* Current involvement in another pain management program or study

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-06-25 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-04 (Estimated)

PRIMARY OUTCOMES:
Pain intensity by The Numeric Pain Rating Scale (NPRS) | Changes in pain intensity at baseline, 6 weeks and 12 weeks.
  The Numeric Pain Rating Scale (NPRS) will be used to assess pain intensity at baseline, 3 weeks, 6 weeks (post-intervention), and 12 weeks (follow-up). Participants will rate their pain on an 11-point scale, ranging from 0 (no pain) to 10 (worst imaginable pain).
Functional disability by The Fibromyalgia Impact Questionnaire (FIQ) | Changes in FIQ at baseline, 6 weeks and 12 weeks.
  The Fibromyalgia Impact Questionnaire (FIQ) will be used to assess functional disability at baseline, 6 weeks, and 12 weeks. The FIQ is a self-report questionnaire containing 21 items related to physical functioning, work status, depression, anxiety, sleep, pain, stiffness, fatigue, and well-being.
Right/left discrimination ability by Recognize smartphone application | Changes in Right/left discrimination ability at baseline, 6 weeks and 12 weeks.
  Recognize app by NOI will be used to assess right/left discrimination ability at baseline, 6 weeks, and 12 weeks. This test will include a series of right/left discrimination tasks similar to those used in the training program.

SECONDARY OUTCOMES:
Cognitive function by The Montreal Cognitive Assessment (MoCA) | Changes in MoCA at baseline, 6 weeks and 12 weeks.
  The Montreal Cognitive Assessment (MoCA) will be used to assess cognitive function at baseline, 6 weeks, and 12 weeks. The MoCA is a brief screening tool designed to detect mild cognitive impairment and includes tasks related to memory, language, visuospatial skills, attention, and executive function.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Director — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No